CLINICAL TRIAL: NCT04387175
Title: Comparison Between an Intraoral Device and Facial Mask for the Early Treatment of Class III Malocclusion: a Randomized Controlled Trial
Brief Title: Intraoral Device vs Facial Mask for Class III Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Franchi, DDS, PhD, Associate Professsor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LF5
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Class III Malocclusion; Dentofacial Anomalies, Including Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Carriere Motion 3D Class III Appliance (Experimental)
  Interventions: Device: Carriere Motion 3D Class III Appliance
- Facial mask (Active Comparator)
  Interventions: Device: Facial mask

INTERVENTIONS:
Device: Carriere Motion 3D Class III Appliance — The device made of stainless steel consists of a flexible bar with two pads at the end which are bonded bilaterally with composite resin to the lower second deciduous molar or the lower first permanent molar at the rear and the lower deciduous canine at the front. The base on the lower deciduous canine has a hook to which bilaterally elastic latex bands are connected with the vestibular tubes of the cemented bands on the upper deciduous second molars (Force 2 elastics ) or on the first permanent upper molars (Force 1 elastics), on whose palatine surface the a rapid maxillary expander is welded.
  Arms: Carriere Motion 3D Class III Appliance
Device: Facial mask — The facial mask consists of a chin pad and frontal pad connected by a central steel bar. On the central bar there is a horizontal steel bar to which latex elastic bands are attached which develop 14 ounces of force. The elastics are connected to the rapid maxillary expander by means of two hooks welded on the bands of the second upper deciduous molars or the first upper permanent molars.
  Arms: Facial mask

SUMMARY:
The aim of this randomized controlled trail is to compare the efficacy of an intraoral device (the Carriere® Motion 3D™ Class III Appliance) with the facial mask for the early treatemnt of Class III malocclusion. This is a monocentric, parallel, controlled trial with blinded examiner.

ELIGIBILITY:
Inclusion Criteria:

* age between 5 and 8 years
* prepubertal patients (cervical vertebral stage 1 or 2)
* Deciduous, early mixed, and intermediate mixed dentition (the lower deciduous canine should show at least 2/3 of the roots unresorbed)
* Presence of Class III skeletal imbalance (Wits appraisal equal to or smaller than
* 1 mm)

Exclusion Criteria:

* Early root resorption of the lower deciduous canines
* Periodontal disease
* Neurologic diseases
* Nickel allergy
* Patients with cleft lip and palate or craniofacial syndromes
* Patients irradiated in the head and neck area
* Patients who have undergone chemiotherapy or immunosuppresive therapy in the previous 5 years
* Patients unable to be followed for at least 1 year

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2021-01-11 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Wits appraisal | Change in Wits appraisal evaluated on the lateral cephalograms taken at the start and at the end of active treatment (6-10 months)
  Distance between the perpendiculars from points A and B on the maxilla and mandible, respectively, onto the occlusal plane

IPD SHARING:
Plan to Share IPD: No